CLINICAL TRIAL: NCT01596322
Title: Novel Approaches to Monitoring and Utilizing Adherence to HIV Therapy in Uganda
Brief Title: International HIV Antiretroviral Adherence, Resistance and Survival
Acronym: UARTO
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of California, San Francisco (Other); Department of Health and Human Services (U.S. Federal Agency); Mbarara University of Science and Technology (Other); University of British Columbia (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jessica Haberer, MD, Associate Professor, Massachusetts General Hospital
Other Study IDs: UARTO, R01 MH054907
Record Dates: First submitted 2010-04-22; First posted 2012-05-11 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: HIV/AIDS
Keywords: HIV/AIDS in resource limited setting; HIV treatment outcomes in resource limited setting; Adherence to HIV treatment in resource limited setting; ART resistance in resource limited setting
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, buffy coat, saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- UARTO

SUMMARY:
Real-time Wireless Adherence Monitoring to HIV Antiretroviral Therapy in Rural Uganda.

DETAILED DESCRIPTION:
The investigators will study use a novel method of real-time wireless adherence monitoring in one of the best established multi-disciplinary HIV antiretroviral treatment cohorts in rural Africa. The investigators will advance our theoretical understanding of HIV antiretroviral adherence behavior, HIV pathogenesis, and to address the monitoring and prevention of HIV antiretroviral treatment failure. Based on a successful pilot study in rural Uganda and favorable cost-effective estimates, the investigators will deploy the Wisepill real-time wireless adherence monitoring system to objectively monitor adherence in real time. The investigators will determine to what extent social capital mitigates economic barriers to long-term adherence and determine if the pervasive impact of stigma on adherence operates through social capital (Aim 1). The investigators will determine the relationship between missed doses, low-level viremia (between 1 and 50 copies RNA/mL), inflammation, bacterial translocation, suboptimal CD4 response, and mortality (Aim 2). Finally, The investigators will examine the relationship between complex adherence patterns and viral failure to both inform selective viral load monitoring and to lay the foundation for the first-of-kind intervention to prevent viral failure after missed doses, but before viral rebound (Aim 3). The investigators will secure behavioral and biologic data over nine years of potential treatment by recruiting 500 additional people to our existing cohort in Mbarara, Uganda for a total of 750 participants.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive patients over 18 years
* ART naive and initiating therapy at the Mbarara Immune Suppression Syndrome (ISS) Clinic
* Live within 60 kilometers of the clinic
* Women who have received a single dose of nevirapine for prevention of mother to child transmission, but have not received other ART, will be included

Exclusion Criteria:

* Patients who do initiate therapy during the course of the study recruitment
* Patients who decline or are unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV positive adults 18 years and older, who are ART naive and initiating ART at either Mbarara HIV clinic or Mulago HIV clinic in Uganda
Sampling Method: Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2004-09 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Adherence to antiretroviral therapy | real time (up to 7 years)
  Adherence is assessed through a medication event monitoring system which records every time the device is opened (e.g. for pill taking). Before June 2012, this data was stored on the device and downloaded monthly. After June 2012, this data is transmitted through cellular networks to a central server in real time.

SECONDARY OUTCOMES:
Correlates of adherence to antiretroviral therapy | every four months
  Questionnaires are administered to participants regarding factors such as depression, stigma, food insecurity, reproductive health, and economic status.
Biological consequences of adherence (or incomplete adherence) | every four months and during adherence interruptions
  Specimens are collected for immunologic and genetic testing at baseline and every four months, as well as during interruptions in adherence as detected by the real time adherence monitoring system.
Adherence to antiretroviral therapy by self report | every four months
  Participants report their adherence over the previous 3 and 28 days by doses missed and visual analog scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Haberer, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mbarara ISS Clinic, Mulago HIV Clinic, Mbarara, Uganda

REFERENCES:
- [Result] Altice FL, Friedland GH. The era of adherence to HIV therapy. Ann Intern Med. 1998 Sep 15;129(6):503-5. doi: 10.7326/0003-4819-129-6-199809150-00015. No abstract available. PMID 9735090
- [Result] Friedland GH, Williams A. Attaining higher goals in HIV treatment: the central importance of adherence. AIDS. 1999 Sep;13 Suppl 1:S61-72. PMID 10546786
- [Result] Sontag D, Richardson L. Doctors withhold H.I.V. pill regimen from some. N Y Times Web. 1997 Mar 2:1, 35. No abstract available. PMID 11647150
- [Result] Tchetgen E, Kaplan EH, Friedland GH. Public health consequences of screening patients for adherence to highly active antiretroviral therapy. J Acquir Immune Defic Syndr. 2001 Feb 1;26(2):118-29. doi: 10.1097/00042560-200102010-00003. PMID 11242178
- [Result] Wainberg MA, Friedland G. Public health implications of antiretroviral therapy and HIV drug resistance. JAMA. 1998 Jun 24;279(24):1977-83. doi: 10.1001/jama.279.24.1977. PMID 9643862
- [Result] Harries AD, Nyangulu DS, Hargreaves NJ, Kaluwa O, Salaniponi FM. Preventing antiretroviral anarchy in sub-Saharan Africa. Lancet. 2001 Aug 4;358(9279):410-4. doi: 10.1016/s0140-6736(01)05551-9. PMID 11502341
- [Result] Popp D, Fisher JD. First, do no harm: a call for emphasizing adherence and HIV prevention interventions in active antiretroviral therapy programs in the developing world. AIDS. 2002 Mar 8;16(4):676-8. doi: 10.1097/00002030-200203080-00025. No abstract available. PMID 11873017
- [Result] UNAIDS. Report on the global HIV/AIDS epidemic. Geneva: UNAIDS, 2002
- [Derived] Chang JL, Tsai AC, Musinguzi N, Haberer JE, Boum Y, Muzoora C, Bwana M, Martin JN, Hunt PW, Bangsberg DR, Siedner MJ. Depression and Suicidal Ideation Among HIV-Infected Adults Receiving Efavirenz Versus Nevirapine in Uganda: A Prospective Cohort Study. Ann Intern Med. 2018 Aug 7;169(3):146-155. doi: 10.7326/M17-2252. Epub 2018 Jun 26. PMID 29946683